CLINICAL TRIAL: NCT05461105
Title: ALTITUDE NASH: A Phase 2, Randomized, Multi-Center, Open-Label Study to Evaluate the Safety and Efficacy of Rencofilstat in Adult Subjects With Nonalcoholic Steatohepatitis Stage 3 Fibrosis
Brief Title: A Study to Evaluate the Safety and Efficacy of Rencofilstat in Adult Subjects With NASH F3
Acronym: ALTITUDE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hepion Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPA-CRV431-210
Record Dates: First submitted 2022-07-13; First posted 2022-07-15 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: NASH With Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: rencofilstat 75 mg (Experimental): 1 rencofilstat 75 mg softgel capsule, 75 mg daily dose, QD 120 days
  Interventions: Drug: rencofilstat, 75 mg
- Cohort B: rencofilstat 150 mg (Experimental): 2 rencofilstat 75 mg softgel capsules, 150 mg daily dose, QD 120 days
  Interventions: Drug: rencofilstat, 150mg
- Cohort C: rencofilstat 225 mg (Experimental): 3 rencofilstat 75 mg softgel capsules, 225 mg daily dose, QD 120 days
  Interventions: Drug: rencofilstat, 225 mg

INTERVENTIONS:
Drug: rencofilstat, 75 mg — 1 softgel capsule
  Arms: Cohort A: rencofilstat 75 mg
Drug: rencofilstat, 150mg — 2 softgel capsules
  Arms: Cohort B: rencofilstat 150 mg
Drug: rencofilstat, 225 mg — 3 softgel capsules
  Arms: Cohort C: rencofilstat 225 mg

SUMMARY:
This is a randomized, open-label, parallel-dosing, multi-center study to evaluate the safety and efficacy of rencofilstat as evidenced by assessing changes in the HepQuant Shunt Disease Severity Index Score (DSI), safety labs, and clinical events in adult NASH subjects with compensated Fibrosis stage F 2/3. Antifibrotic biomarker activity will be evaluated on an exploratory basis.

DETAILED DESCRIPTION:
This study consists of 3 phases: (i) Screening and Randomization; (ii) treatment; and (iii) follow up. During Screening, each subject will provide informed consent prior to starting any study specific procedures. The randomization of the NASH F3 subjects will be performed in a 1:1:1 ratio between rencofilstat 75 mg, rencofilstat 150 mg, and rencofilstat 225 mg. During the treatment period, randomized subjects will be provided the treatment and assessments to monitor safety, tolerability and efficacy. All subjects will receive study drug in the morning. Prior to dosing, subjects can have a light breakfast, avoiding high fat meals. In the follow up phase, investigational product (IP) will be discontinued followed by 14 days of safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between 18 and 75 years of age (inclusive).
2. BMI above 25.0 kg/m2
3. Biopsy confirmed NASH with histologic liver fibrosis stage 3 as defined by the Nonalcoholic Steatohepatitis Clinical Research Network (NASH CRN) scoring of liver fibrosis based on available historical biopsy report if the following are met:

   i. Historical biopsy was obtained no more than 6 months (180 ± 5 days) prior to the first day of Screening. ii. No new therapeutic intervention for NASH of at least 2 or more weeks was made during the preceding 3-month (90-day) period (e.g., vitamin E ≥ 400 IU/day, pioglitazone, or incretins [e.g., liraglutide, semaglutide]). Subjects may be treated with vitamin E or pioglitazone as long as such subjects are maintained on a stable dose for 3 months prior to randomization, and the dose should be held constant during the trial.
4. Subjects without historical biopsy will be eligible for inclusion if their AGILE 3+ score using the FibroScan Diagnostic App is ≥0.53. The AGILE 3+ score is composed of: FibroScan fibrosis score, laboratory values (AST, ALT, Platelets), and clinical parameters (Age, Sex, Diabetes status) to calculate the AGILE 3+ score.

Exclusion Criteria:

1. Positive test for hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or human immunodeficiency virus antibodies (HIVAb). If HCVAb test is positive, then an HCV-RNA test will be performed. If this test is negative, the subject is allowed to participate in the study, as long as the subject meets all other inclusion criteria and has never been treated for HCV or was treated >2 years ago and achieved a sustained virologic response at that time.
2. Subjects with symptomatic severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) infection identified during the screening period.
3. At screening, subjects with uncontrolled hypertension (either treated or untreated) defined as a systolic blood pressure >160mmHg or a diastolic blood pressure of >110mmHG.
4. Subjects on either a non-selective beta blocker or an angiotensin-converting enzyme (ACE) inhibitor or angiotensin II receptor blocker (ARB) who are unwilling/unable to delay taking their normal dose the morning of HepQuant testing.
5. Subjects with transaminases >5 x upper limit of normal (ULN).
6. Subjects with ALP >2 x ULN.
7. Subjects with total serum bilirubin >1.5 x ULN, unless the subject has Gilbert's Syndrome, in which case the subject can be enrolled provided the direct bilirubin is within 30% of the total bilirubin.
8. Subjects with a platelet count <140,000/mm3.
9. Subjects with an INR ≥ 1.3 in the absence of anticoagulants.
10. Subjects with albumin <3.5 g/dL.
11. Model for End-Stage Liver Disease (MELD) score >12, unless due to an alternate etiology such as therapeutic anticoagulation or Gilbert's.
12. An estimated glomerular filtration rate (eGFR) <60 mL/min/1.73 m2 (calculated by the Chronic Kidney Disease Epidemiology Collaboration [CKD-EPI] method).
13. Subjects with hemoglobin A1c (HbA1c) >9.5%.
14. Other well documented causes of chronic liver disease according to standard diagnostic procedures.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-03-15 (Actual); Primary Completion 2023-04-15 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline in DSI score of subjects taking rencofilstat (75 mg, 150 mg, 225 mg), determined using HepQuant SHUNT Test, on Day 60, and Day 120. | 120 Days
  Primary Efficacy Endpoint
The percent of subjects taking rencofilstat (75 mg, 150 mg, 225 mg) that have experienced treatment-emergent adverse events, serious adverse events, adverse events of special interest, physical and laboratory abnormalities. | 120 Days
  Primary Safety Endpoint

CONTACTS AND LOCATIONS:
Locations (20):
- United States (20):
  - Arizona Liver Health-Chandler, Chandler, Arizona
  - Arizona Liver Health-Glendale, Peoria, Arizona
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Arizona Liver Health-Tucson, Tucson, Arizona
  - Velocity Clinical Research-Chula Vista, Chula Vista, California
  - Velocity Clinical Research-San Diego, La Mesa, California
  - Synergy Healthcare, LLC, Bradenton, Florida
  - Covenant Metabolic Specialists-Fort Myers, Fort Myers, Florida
  - Evolution Clinical Trials, Inc., Hialeah Gardens, Florida
  - Progressive Medical Research, Port Orange, Florida
  - Covenant Metabolic Specialists-Sarasota, Sarasota, Florida
  - Clinical Research Institute of Michigan, Chesterfield, Michigan
  - Coastal Reseach Institute, Fayetteville, North Carolina
  - Optimed Research, Columbus, Ohio
  - Clinical Research Institute of Ohio, Westlake, Ohio
  - Pinnacle Clinical Research-Austin, Austin, Texas
  - Apex Mobile Clinical Research, Bellaire, Texas
  - South Texas Research Institute, Edinburg, Texas
  - Pinnacle Clinical Research-Georgetown, Georgetown, Texas
  - Pinnacle Clinical Research-San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Mayo P, Hobbs T, Zhao C, Canizares C, Foster R, McRae MP, Helmke SM, Everson GT. Rencofilstat Treatment Improves Liver Function in MASH With Advanced Fibrosis as Quantified by HepQuant DuO. Liver Int. 2025 Mar;45(3):e70036. doi: 10.1111/liv.70036. PMID 39982177